CLINICAL TRIAL: NCT00187746
Title: Effect of Age on the Renal Clearance of Adefovir
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Budget exceeded for project.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 992
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Other Conditions That May Be A Focus of Clinical Attention
Keywords: Healthy Control
MeSH Terms: interventions — adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Age 18-25 years (Experimental): African American subjects between the ages 18 to 25 years given Adefovir dipivoxil.
  Interventions: Drug: Adefovir dipivoxil
- Age 48-55 years (Experimental): African American subject between the ages 48 to 55 years given Adefovir dipivoxil.
  Interventions: Drug: Adefovir dipivoxil

INTERVENTIONS:
Drug: Adefovir dipivoxil — Subjects will be given a single oral dose of 10 mg of adefovir dipivoxil
  Other Names: HEPSERA® is the tradename

SUMMARY:
Healthy African American subjects with normal hepatic and renal function will be administered 10mg adefovir dipivoxil in a fasting state. Subjects will have blood and urine collections over the following 24 hours for the measurement of adefovir renal clearance. To investigate the role of age in renal adefovir elimination, 8 subjects will be enrolled from each of the following age groups: 18-25 years and 48-55 years.

DETAILED DESCRIPTION:
There are two major routes of elimination for drugs - hepatic metabolism and renal elimination. For small, hydrophilic molecules, the renal route predominates. The renal function of patients taking these medications therefore determines the pharmacokinetics of (and by extension the clinical response to) these medications. One of the most common causes of reduced renal function is a decline with age.

Renal drug elimination is comprised of passive drug filtration, active secretion, and reabsorption (which can occur by both active and passive processes). The filtration function of the kidney, approximated by the glomerular filtration rate (GFR) falls by 25-50% between the ages of 20 and 90 [Turnheim 2003]. The decline in renal function with age has been identified as a major cause of adverse drug reactions in the elderly population [Lindeman 1995; Mühlberg 1999]. To avoid overdosing and exaggerated responses from these medications, algorithms have been established for dosing in patients with reduced renal function due to changes in glomerular filtration.

However, in a previous study looking at the pharmacokinetics of a drug cleared only by the renal route, we made an observation that appeared to contradict the "renal clearance declines with age" dogma. In this study, Effect of Genetic Variation in the Renal Transporter, OAT1, on the Renal Secretion of Adefovir), we identified individuals with genetic variants in OAT1, a transporter that was believed to be involved in the active secretion of Adefovir. All OAT1 non-synonymous genetic variants we identified were in the African American population. We administered 10mg Adefovir dipivoxil to 10 African American subjects between the ages of 19 and 49 (4 who had a genetic variant in OAT1, and six without one). These subjects were identified from a parent study, called "SOPHIE" (NCT00187668). SOPHIE (Studies Of Pharmacogenetics In Ethnically Diverse Individuals) is a study where DNA was collected from Bay Area adults (18-40 years of age) for the testing of drug response genes. In addition to DNA donation, subjects consent to be contacted for future studies.

We collected blood and urine over 24 hours to calculate the total renal clearance and net secretory clearance of adefovir. Although we saw no difference in the renal elimination of adefovir in the subjects attributable to OAT1 variants, we found a correlation between the age and renal clearance. Filtration (calculated from the measured creatinine clearance) remained constant in this population (112 ml/min + 18 (SD)), and the clearance of Adefovir increased with age. Both the total renal clearance and net secretory clearance increased with age (p=0.017 and p=0.010, respectively).

This incidental finding is interesting, as it may indicate an age-dependence of active drug elimination mechanisms. However, the sample size in this previous study is small, and the observation may not be accurate. We therefore have planned this confirmatory study, to expand the study population. As the initial finding was made in African American subjects, we plan to enroll an additional 16 African American subjects (8 each from the following age groups: 18-25 and 48-55). We will also genotype these individuals for variants in transporters and other proteins that may play a role in adefovir renal elimination. If the unexpected finding of an age-related increase of adefovir renal clearance is observed in this study, additional follow-up studies will be planned to examine whether the same holds true for other ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

1. African American (either male or female);
2. Between the ages of 18 and 25 OR between the ages of 48 and 55;
3. Healthy (no self-reported ongoing medical conditions, and no clinically significant laboratory findings from a CBC and Complete Metabolic Panel);
4. Willing to participate in the study.

Exclusion Criteria:

1. Subject has a medical condition that increases the risks of study participation (including pregnancy and poor renal function as defined by a calculated ClCr < 60 ml/min);
2. Any subjects with a laboratory value out of normal range and deemed to be potentially clinically significant will be excluded. Specifically, individuals with anemia (hemoglobin < 12 g/dL) or an elevation in liver enzymes (alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, glutamyltransferase) to higher than double the respective normal value will be excluded;
3. Subject is taking any medication other than vitamins or oral contraception;
4. Subject does not consent to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Renal Clearance of adefovir | 24 hours
  To investigate the role of age in renal adefovir elimination, 8 subjects will be enrolled from each of the following age groups: 18-25 years and 48-55 years.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Giacomini, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Fujita T, Brown C, Carlson EJ, Taylor T, de la Cruz M, Johns SJ, Stryke D, Kawamoto M, Fujita K, Castro R, Chen CW, Lin ET, Brett CM, Burchard EG, Ferrin TE, Huang CC, Leabman MK, Giacomini KM. Functional analysis of polymorphisms in the organic anion transporter, SLC22A6 (OAT1). Pharmacogenet Genomics. 2005 Apr;15(4):201-9. doi: 10.1097/01213011-200504000-00003. PMID 15864112